CLINICAL TRIAL: NCT06034938
Title: DOR/TDF/3TC Maintenance Therapy Among Patients Harboring M184V/I Mutation: a Pilot Open-label Study
Brief Title: DOR/TDF/3TC Switch With M184V/I in People With Controlled HIV (Drive Off-Road)
Acronym: DOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP-RC_Parienti007
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hiv
Keywords: doravirine; M184 mutation; Maintenance therapy; PLWH
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — doravirine; Lamivudine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative, single arm pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm DOR/3TC/TDF (Experimental): Doravirine 100 mg Lamivudine 300 mg Tenofovir disoproxil fumarate 245 mg Delstrigo (R): 1 pill/day for 48 weeks
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate 100 MG-300 MG-300 MG Oral Tablet [DELSTRIGO]

INTERVENTIONS:
Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate 100 MG-300 MG-300 MG Oral Tablet [DELSTRIGO] — Switch previous therapy with DOR/TDF/3TC
  Other Names: Delstrigo

SUMMARY:
The goal of this pilot, phase 2, single-arm, clinical trial is to assess the antiretroviral combination Doravirine (DOR)/Lamivudine (3TC)/Tenofovir Disproxyl Fumarate (TDF) in participants with suppressed HIV who previously developed M184V/I mutation that confers resistance to 3TC. The main question it aims to answer is to explore the rate of HIV suppression 24 weeks after the switch to DOR/3TC/TDF. The study follow-up will continue until 48 weeks. Other endpoints will be metabolic changes, weight changes, modification in the HIV-DNA mutations overtime. Eligible participants will switch from their prior regimen to DOR/3TC/TDF with careful HIV-RNA monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult living with HIV
* Receiving stable antiretroviral treatment for at least 3 months
* HIV RNA VL<50cp/mL for at least 6 months
* Presence of the M184V/I mutation in at least one previous genotype performed on plasma HIV RNA but absent from the genotype on current standard pro-viral DNA (Sanger technique)
* Signed informed consent

Exclusion Criteria:

* History of genotypic mutation associated with resistance to DOR or TDF according to the ANRS version 32 algorithm, i.e. :
* For DOR : V106A/M; Y188L; G190E/S; M230L; L100I + K103N; K103N + Y181C; K103N + P225H; F227C; At least 3 amongst: A98G, L100I, K101E, V106I, E138K, Y181C/V, G190A or H221Y
* For TDF : At least 3 mutations among: M41L, E44D, D67N, T69D/N/S, L74V/I, L210W, T215A/C/D/E/G/H/I/L/N/S/V/Y/F; K65R/E/N ; Insertion at codon 69; K70E
* Contraindications to the use of DOR/TDF/3TC
* Hypersensitivity to doravirine, tenofovir, lamivudine or any of the excipients (lactose in particular)
* Current or recent treatment with a strong CYP3A4 inducer
* Breast-feeding
* Patients already on DOR
* Pregnant or breast-feeding women
* Patients under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Plasma HIV-RNA at 24-week | 24 weeks from the switch to DOR/3TC/TDF
  Number of copies/mL

SECONDARY OUTCOMES:
Plasma HIV-RNA at 48-week | 48 weeks from the switch to DOR/3TC/TDF
  Number of copies/mL

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Caen, Caen
  - CHU Orléans, Orléans
  - CHU Rouen, Rouen
  - CH Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: Yes
Contact principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2-year after publishing the princeps study
Access Criteria: Relevant scientific question with protocol